CLINICAL TRIAL: NCT00624728
Title: Assessment of 18Fluoro-thymidine PET-CT for the Volume Definition of High-grade Gliomas (GLIO-TEP) : Correlation With Histopathology
Brief Title: Assessment of 18FLT PET-CT for Volume Definition of High-grade Gliomas (GLIO-TEP)
Acronym: GLIO-TEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9420-04; 2004-033
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: High-grade Glioma; Astrocytoma; Glioblastoma
Keywords: Positron-Emission Tomography; Alovudine [Substance Name]; 18F-FLT; Magnetic Resonance Imaging; Astrocytoma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Radiation: 18F Fluorothymidine PET CT

INTERVENTIONS:
Radiation: 18F Fluorothymidine PET CT — 18 FLT will be provided by the Laboratoire des Radiopharmaceutiques- Université Bordeaux2, Hôpital Xavier Arnozan and prepared according to the method described by Grierson and Shields ( Grierson J, Shields A. Nucl Med Biol 27 :143-156 ; 2000).
  Specific activity of 18FLT will be more than 37 GBq/µmol (>1Ci/µmol) corrected for decay at the end of bombardment of cyclotron target. Before tracer injection to patients, each dosis will be tested for pH and for radiochemical purity (> 95%) via HPLC technique and thin layer chromatography.
  18FLT dosis will be injected intravenously to the patients (10 mL of salted isotonic solution with less than 10 % (v/v) of ethanol (USP). Administrated activity will be calculated estimating total body surface of patient (2,6 MBq/kg ou 0,07 mCi/kg) with maximal activity of 185 MBq.
  PET acquisition will be realized as follows : Dynamic acquisition in 3D mode for 35 min, Iterative reconstruction (OSEM) with and without attenuation correction.

SUMMARY:
18F-Fluorothymidine is a recently developed PET tracer to image tumor cell proliferation. Very few data report an interest of using such a tracer for cerebral malignant tumor management. In our project, we want to compare the tumoral volumes obtained with PET and MRI, with the gold standard histopathological diagnosis according to the WHO grading malignancy scale and the Ki-67 proliferation index, for preoperative evaluation as much as for tumoral postoperative residue evaluation. Furthermore, we want to explore the interest of 18F-FLT-PET volume to better delineate tumoral volume in radiotherapeutic management of gliomas.

DETAILED DESCRIPTION:
* Background: 18FDG is the most widely used tracer for oncologic positron emission tomography (PET). However, the high glucose utilization of normal gray matter limits its utility in brain explorations. More recently, 18FLT was introduced as a PET tracer for tumor imaging. It has been found useful for non-invasive assessment of the proliferation status of various tumors. Its potential clinical use in the evaluation of brain tumors has not been clearly determined because of sparse studies.
* The primary objective of this study is to assess the positive predictive value of PET-CT uptake of 18FLT in diagnosing malignant tissue by comparison with the histopathological gold standard diagnosis according to the WHO grading malignancy scale and the Ki-67 proliferation index, at the time of preoperative evaluation.
* Secondary objectives are: to describe and compare preoperative tumor volumes and postoperative residual tumor volumes as assessed by 18FLT PET-CT and MRI, and to describe a quantitative proliferation index with PET (SUV for "standardized uptake value").
* Study design: This is an exploratory cross-sectional study at two separate times: pre-and postoperative. Eligible patients will be included consecutively. Histological samples will be analyzed blindly to imaging data. Assessments of PET-CT and MRI volumes will be blind to each other.
* Procedure: After information and written informed consent and before surgery, patients will undergo MRI and 18F-FLT PET-CT to obtain the tumor volume according to both modalities. Then, surgeons will make different biopsies from i) areas with MR abnormalities and FLT uptake, ii) area with FLT uptake and no MR abnormality (on the surgery approach way or in not functional areas), iii) area with MR abnormality without any FLT uptake, iiii) area without any uptake where biopsy is possible because the area is on the surgery approach way. Then, the samples will be blindly analyzed to determine the Ki-67 proliferation index and WHO grading malignancy scale. Patients will undergo again 18F-FLT PET-TDM and MRI at least 4 weeks after surgery, in the week preceding radiotherapy, to determine residual tumor volumes.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18
* suspicion of malignant glioma on MRI aspect
* surgical indication with neuronavigation
* signed informed consent
* absence of contraindication for MRI
* absence of pregnancy or breast-feeding

Exclusion Criteria:

* women : pregnancy or breast-feeding or no oral or intra-uterine contraception (if not post-menopause)
* secondary exclusion if high grade glioma diagnostic (glioblastoma or astrocytoma grade III) is not confirmed after surgery with histopathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Predictive positive value of PET uptake for detection of malignant tissue (defined with Ki-67 proliferation index >15% in PET+ volumes) | before and during surgery

SECONDARY OUTCOMES:
Comparison of volumes defined by PET and MRI | before surgery and 4 weeks after surgery
Description of a quantitative PET proliferation index ("standardized uptake value") | before surgery and 4 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez Philippe, Dr, Principal Investigator — University Hospital, Bordeaux, France; Perez Paul, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (2):
- France (2):
  - Hôpital St André, CHU de Bordeaux, Bordeaux
  - Hôpital Pellegrin-tripode , CHU de Bordeaux, Bordeaux

REFERENCES:
- [Background] Choi SJ, Kim JS, Kim JH, Oh SJ, Lee JG, Kim CJ, Ra YS, Yeo JS, Ryu JS, Moon DH. [18F]3'-deoxy-3'-fluorothymidine PET for the diagnosis and grading of brain tumors. Eur J Nucl Med Mol Imaging. 2005 Jun;32(6):653-9. doi: 10.1007/s00259-004-1742-3. Epub 2005 Feb 15. PMID 15711980
- [Background] Chen W, Cloughesy T, Kamdar N, Satyamurthy N, Bergsneider M, Liau L, Mischel P, Czernin J, Phelps ME, Silverman DH. Imaging proliferation in brain tumors with 18F-FLT PET: comparison with 18F-FDG. J Nucl Med. 2005 Jun;46(6):945-52. PMID 15937304